CLINICAL TRIAL: NCT06789900
Title: Targeting mTOR With Everolimus and/or Physical Training for Preventing Postmenopausal Bone Loss and Accelerated Skeletal Aging: The RapaLoad Study
Brief Title: Everolimus and/or Exercise to Prevent Bone Loss in Postmenopausal Women
Acronym: RapaLoad
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark. (Unknown); OPEN - Odense Patient data Explorative Network, The University of Southern Denmark, Odense, Denmark (Unknown); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EU CT: 2023-508093-28-00
Record Dates: First submitted 2024-11-27; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Women
Keywords: Everolimus; Exercise; Football training session; postmenopausal women; bone loss; skeletal aging
MeSH Terms: conditions — Motor Activity; Bone Diseases, Metabolic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): Participants will be asked to continue their life as usual with no specific recommendation
- Football fitness group (Experimental): Participants will join structured hybrid exercise training via the "football fitness concept" designed for participants with little prior experience with football and it is multifaceted training incorporating endurance training, high-intensity interval training (HIIT) and strength training. The training session lasts 60 minutes, and participants will receive two training sessions per week for 24 weeks. Each session is composed of: a 15 min warm-up that includes strength and balance exercises, a 15 min period with technical pair-based drills, and a 30-min period with small-sided football drills.
  Interventions: Other: Football Fitness Concept
- Everolimus group (Experimental): Participants will take an oral dose of everolimus 5 mg once a week for 24 weeks.
  Interventions: Drug: Everolimus (Afinitor®)
- Everolimus and Football fitness group (Experimental): Participants will join structured hybrid exercise training via the "football fitness concept" designed for participants with little prior experience with football and it is multifaceted training incorporating endurance training, high-intensity interval training (HIIT) and strength training. The training session lasts 60 minutes, and participants will receive two training sessions per week for 24 weeks. Each session is composed of: a 15 min warm-up that includes strength and balance exercises, a 15 min period with technical pair-based drills, and a 30-min period with small-sided football drills and take an oral dose of everolimus 5 mg once a week for 24 weeks.
  Interventions: Drug: Everolimus (Afinitor®); Other: Football Fitness Concept

INTERVENTIONS:
Drug: Everolimus (Afinitor®) — Oral dose of everolimus 5 mg once a week for 24 weeks
  Other Names: Football fitness session
  Arms: Everolimus and Football fitness group; Everolimus group
Other: Football Fitness Concept — Structured hybrid exercise training via the "football fitness concept" organized as a super-vised group training at the University of Southern Denmark, Department of Sports Science and Clinical Biomechanics. "Football Fitness concept" is designed for participants with little prior experience with football and it is multifaceted training incorporating endurance training, high-intensity interval training (HIIT) and strength training. The training session lasts 60 minutes, and participants will receive two training sessions per week for 24 weeks. Each session is composed of 4 elements: a 15 min warm-up that includes strength and balance exercises, a 15 min period with technical pair-based drills, and a 30-min period with small-sided football drills
  Arms: Everolimus and Football fitness group; Football fitness group

SUMMARY:
It is estimated that women lose around 20-25% of bone mass during the 5-10 years period of postmenopausal transition, and menopause is considered a major risk factor for osteoporotic fragility fracture. Currently, there is no preventive strategy to counteract these changes, and hormone replacement therapy is not considered an attractive option for many women, because of concerns related to side effects. Rapamycin, through inhibition of mTOR (the mechanistic target of Rapamycin) has been demonstrated in many preclinical animal models to extend lifespan and healthspan. The most well-established mTOR inhibitors include rapamycin (sirolimus) and its analog (also referred as rapalog). Everolimus are FDA approved and have been used for many years at a high dose as an immunosuppressant and anti-cancer drug. Exercise training has been demonstrated to counteract age-related degenerative changes in several clinical studies. The aim of this randomized clinical trial is to test the effects of treatment with oral Everolimus, exercise, or their combination as a preventive strategy for impaired musculoskeletal function in healthy postmenopausal women.

The trial will include 136 women aged 45-60 years with T-score >-3 and no history of hip, Colles' or symptomatic vertebral fractures within the last 6 months, randomized to 24 weeks of treatment with one of the following regimens:

1. control group getting general health advice,
2. Football fitness session group, physical training consisting of structured hybrid exercise training via the "football fitness concept" for 1hour, 2 times/ week
3. Everolimus group receiving an oral dosage of 5 mg everolimus once a week, (4) Everolimus and football fitness session group, consisting of structured hybrid exercise training via the "football fitness concept" for 1 hour, 2 times/week combined with oral everolimus 5 mg once a week.

The primary outcome of this trial is percentage change in bone formation marker P1NP (Procollagen Type 1 propeptide) between baseline and week 24. Secondary outcomes include percentage changes in bone resorption marker CTX (cross-lined C-telopeptide of type 1 collagen), bone mineral density (BMD), bone structure as determined by high resolution CT-scanning, muscle function and postural balance. As exploratory endpoints, changes in biological age as determined by "epigenetic clocks", levels of senescence-associated secretory phenotype (SASP) as an indicator of whole-body burden of senescent cells.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 45-60 years old as evidenced by measuring serum levels of LH and FSH and absence of menstruation for at least 1 year.
* No history of low energy hip or vertebral fractures during the last 6 months.
* Ability to provide informed consent.

Exclusion Criteria:

* Diabetes (type 1 and 2)
* Heart failure similar to NYHA Class IV
* Primary hyperparathyroidism
* Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, severe renal impairment (eGFR <20) or liver function (baseline phosphatase higher than twice upper limit (105 U/L)), active rheumatic diseases, celiac disease, severe chronic obstructive lung disease (COPD), hypopituitarism, or Cushing's disease.
* Previous use of bone antiresorptive or bone anabolic drugs within the last 5 years.
* Use of anabolic steroids in the previous year
* Treatment with drugs known to affect cytochrome P450 3A due to its role in everolimus metabolism
* History of coagulopathy or medical condition requiring long-term anticoagulation
* Anemia - Hg < 9.0 g/dl, Leukopenia - white blood cells (WBC) < 3,500/mm3, Neutropenia absolute neutrophil count < 2,000/mm3, or Platelet count - platelet count < 125,000/mm3
* Patients with impaired wound healing or history of a chronic open wound
* Scheduled for immunosuppressant therapy for transplant or scheduled to undergo chemotherapy or any other treatment for malignancy
* Untreated dyslipidemia with LDL-c > 4.9 mmol/L and family history of dyslipidemia, Total cholesterol > 9.1 mmol/L, or triglycerides > 9.9 mmol/L
* Any form of clinically relevant primary or secondary immune dysfunction or deficiency
* Unstable ischemic heart disease
* Bone mineral density (BMD) measured by DXA scanning with T-score <-3
* Known allergy to rapamycin or rapalogs
* The study will exclude participants with inability to speak and understand Danish and with inability to cooperate or perform physical training.
* Inability to give informed consent

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 136 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Procollagen type 1 N-terminal propeptide (P1NP) | Baseline and 24 weeks
  Percentage change in circulating levels of bone formation marker N-terminal fragment of procollagen type 1 (P1NP) at 24 weeks as compared with baseline

SECONDARY OUTCOMES:
Bone resorption markers (CTX and TRAcP) | Baseline, week 2, week 4, week 12 and week 24
  Change in circulating levels of bone resorption markers (C-terminal telopeptide of type 1 collagen (CTX) and Tartrate resistant acid phosphatase (TRAcP))
Bone formation markers (Osteocalcin, bALP, P1NP (other time points)) | Baseline, week 2, week 4, week 12 and week 24 (P1NP: week 2, week 4 and week 12)
  Change in circulating levels of bone formation markers (osteocalcin, and bone alkaline phosphatase) and additional time point for P1NP
Bone mineral density (BMD) | Baseline, week 24
  Lumbar spine (L1-4), and total hip and femoral neck bone mineral density (BMD) measured by dual-energy X-ray absorptiometry (DXA)
Bone microarchitecture, mass and geometry | Baseline, week 24
  Bone microarchitecture at the distal radius and tibia assessed using high-resolution peripheral quantitative computed tomography (HR-pQCT)
Muscle fitness and postural balances (test 1) | Baseline, week 24
  Y-balance test
Muscle Fitness and postural balances (test 2) | Baseline, week 24
  Stork balance test
Muscle fitness and postural balances (test 3) | Baseline, week 24
  Handgrip strength test
Muscle fitness and postural balances (test 4) | Baseline, week 24
  leg strength test- knee extension and knee flexion tests
Muscle fitness and postural balances (test 5) | Baseline, 24 weeks
  Sit-to-stand chair test
Muscle fitness and postural balances (test 6) | Baseline, week 24
  stair climb test
Muscle fitness and postural balances (test 7) | Baseline, week24
  Counter Movement Jump test
Cardiopulmonary health (test 1) | Baseline, week 24
  Vo2 max (seismofit)
Cardiopulmonary health (test 2) | Baseline, week 24
  Bicycle test with submaximal exercise (warm-up, submax HR and fat oxidation)
Cardiopulmonary health (test 3) | Baseline, 24 weeks
  5-s peak power test
Cardiopulmonary health (test 4) | Baseline, week 24
  maximal oxygen uptake test
Cardiopulmonary health (test 5) | Baseline, week 24
  6-min walk test
Metabolic health (test 1) | Baseline, week 24
  weight, lean and fat body mass by DXA scanning
Metabolic health (test 2) | Baseline, week 24
  Fasting blood glucose
Metabolic health (test 3) | Baseline, week 24
  Fasting insulin
Metabolic health (test 4) | Baseline, week 24
  Lipid parameters

OTHER OUTCOMES:
SF-12 | Baseline, week 24
  Quality of life questionnaire
SASP | Baseline, week 24
  Serum levels of senescence associated secretory phenotype (SASP), which reflect the whole-body burden of senescent cells

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Kassem, DMSc, PhD, Principal Investigator — Odense University Hospital; Florence Figeac, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
After completion of the project and irrespective of the outcomes, de-identified trial results will be published in peer-reviewed journals and www.clinicaltrials.gov. A summary of the clinical trial results will be presented in a language understandable to the layperson and made available in the EU database.